CLINICAL TRIAL: NCT06465381
Title: Safety Planning and Cognitive Behavioral Therapy for Adolescent Suicide Prevention in Mozambique: A Hybrid Effectiveness/Implementation Cluster Randomized Trial
Brief Title: Safety Planning and Cognitive Behavioral Therapy for Adolescent Suicide Prevention in Mozambique
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Bradley Wagenaar, Associate Professor, Global Health, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00019158; R01MH134882 (NIH)
Record Dates: First submitted 2024-06-11; First posted 2024-06-18 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Suicide Prevention
Keywords: Suicidal Behavior; Safety Planning Intervention; Transdiagnostic Cognitive Behavioral Therapy for Suicide Prevention; Suicidal Ideation; Depressive Symptoms
MeSH Terms: conditions — Suicide Prevention; Suicidal Ideation; Depression

STUDY DESIGN:
Intervention Model Description: Using a three-arm parallel cluster RCT the investigators will randomize 7 secondary schools each to enhanced usual care, Safety Planning Intervention, and Transdiagnostic Cognitive Behavioral Therapy for Suicide prevention (21 schools total) to evaluate effects on suicidal behaviors (primary) and suicidal ideation/depressive symptoms (secondary). EUC will involve screening and active referral to government youth friendly mental health service programs.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Enhanced Usual Care (Other): In school randomized to EUC, youth who are determined to be high risk of suicide using the C-SSRS will be transported to the local government emergency psychiatric services that Dr. Cumbe (Co-I) directs in his role as Provincial Director of Mental Health services in Sofala Province. For students with moderate risk, they will receive information and referral to local government mental health and youth friendly services. At follow-up outcome ascertainment time points, those in the EUC arm will be re-assessed for suicide risk and uptake of referral services.
  Interventions: Behavioral: Enhanced Usual Care
- Safety Planning Intervention (Experimental): If the student attends a school that has been randomized to SPI alone, youth will be asked to participate in a collaborative approach to create a stepwise safety plan that includes a simple list of individually tailored, concrete coping mechanisms to be enacted during or leading up to a crisis. The seven steps of the safety plan include: 1) recognizing warning signs of a crisis; 2) employing internal coping strategies; 3) using social contacts and settings to distract from suicidal thoughts; 4) seeking help from family members or close friends; 5) contacting healthcare or emergency services; and 6) reducing access to means. Youth will be followed-up at 2- and 4-weeks post intake to assess suicide risk and review their safety plan. Youth who are determined to be high risk of suicide using the C-SSRS will be transported to the local government emergency psychiatric services.
  Interventions: Behavioral: Safety Planning Intervention
- Transdiagnostic Cognitive Behavioral Therapy for Suicide Prevention (Experimental): In schools randomized to TCBT-S, youth will receive 1) the safety planning intervention as outlined above 2) psychoeducation focused on suicidal thoughts and behaviors and how TCBT-S is expected to contribute to recovery; 3) cognitive restructuring adapted to focus on the thoughts and feelings that occur during individual's suicidal thoughts or behaviors; 4) linking the getting active module to coping strategies included in the safety plan for acute distress tolerance and crisis avoidance; and 5) problem solving focused on addressing problems believed to be contributing to suicidal thoughts and behaviors; and 6) relaxation techniques to help manage overwhelming emotions and/or physical sensations that may contribute to suicidal thoughts and behaviors. TCBT-S will be implemented in 6-8 sessions each spaced one week apart. Youth who are determined to be high risk of suicide using the C-SSRS will be transported to the local government emergency psychiatric services.
  Interventions: Behavioral: Transdiagnostic Cognitive Behavioral Therapy for Suicide Prevention

INTERVENTIONS:
Behavioral: Safety Planning Intervention — All behavioral interventions will be provided by a trained nonspecialist healthcare worker, descriptions of each intervention can be found under treatment arm/group descriptions.
  Arms: Safety Planning Intervention
Behavioral: Enhanced Usual Care — All behavioral interventions will be provided by a trained nonspecialist healthcare worker, descriptions of each intervention can be found under treatment arm/group descriptions.
  Arms: Enhanced Usual Care
Behavioral: Transdiagnostic Cognitive Behavioral Therapy for Suicide Prevention — All behavioral interventions will be provided by a trained nonspecialist healthcare worker, descriptions of each intervention can be found under treatment arm/group descriptions.
  Arms: Transdiagnostic Cognitive Behavioral Therapy for Suicide Prevention

SUMMARY:
This implementation research project aims to test the effectiveness and implementation outcomes of suicide safety planning along and a transdiagnostic cognitive behavioral intervention for suicide prevention on decreasing suicidal behaviors in secondary school students in Mozambique. This study will also result in hypothesized mechanisms of intervention effects, costs and cost-effectiveness.

DETAILED DESCRIPTION:
More than 75% of suicide deaths occur in low-and middle-income countries (LMICs) and almost 90% of adolescents who die by suicide live in LMICs. Globally, suicide is the fourth leading cause of death for youth and young adults aged 15-29. The African WHO region has the highest age-standardized suicide rates in the world, with countries like Mozambique having suicide rates almost three times the global average. Six of the top 10 countries by suicide rates in the world are in the African region. Despite this, there are few to no evidence-based adolescent suicide prevention packages developed for, and tested in, the African context. This is an urgent need to safeguard the well-being of youth and young adults.

Data from the investigative team suggest that 15-25% of high school students in Mozambique are experiencing current suicidal ideation (SI), ~40% of those with ideation have past month suicidal behavior (SB), and 9% have had a lifetime suicide attempt. Approximately 50% of youth expressing SI or SB also express clinically significant symptoms of depression, anxiety, and/or PTSD. To address this problem, the proposed work builds upon innovations in the field and a decades-long partnership between the University of Washington and government partners in Mozambique. First, while the Suicide Safety Planning Intervention (SPI) has evidence in high-income contexts, investigators have conducted what the investigators believe to be the first pilot of SPI among adolescents 12-19 in the African region and found it feasible for delivery by non-specialists and acceptable by adolescents. Second, the investigative team adapted and demonstrated the feasibility, acceptability, and initial effectiveness of the Common Elements Treatment Approach (CETA-MZ), a transdiagnostic CBT-based therapy delivered by non-specialists in Mozambique. For young adults aged 18-24, CETA-MZ was shown to decrease depressive symptoms by 80% and reduce suicidal ideation from 20% to <3% by visit five. The results of this work have led to the national scale-up of CETA-MZ in HIV/AIDS settings in Mozambique. The investigators believe that these two evidence-based practices, both with demonstrated feasibility in Mozambique, have the potential to be powerful interventions to prevent adolescent suicidal behavior. Yet, a recent meta-analysis found lower comorbidity of psychiatric disorders and suicidal behavior in LMICs (~50%) compared to high-income countries (~90%). Therefore, it is possible that applying CETA-MZ to address psychiatric symptoms may not lead to significant decreases in suicidal behavior above and beyond SPI alone. For these reasons, the investigators propose to test both SPI alone and the integration of SPI into CETA-MZ - adapted for adolescent suicide prevention - to create a transdiagnostic CBT intervention for suicide (TCBT-S) delivered by non-specialists in Mozambican secondary schools. Due to limited resources for mental health in the African region the investigators aim to test whether the potential gains in effectiveness with the more resource intensive TCBT-S justify its scale-up versus the brief SPI intervention. This study will also generate evidence on costs, implementation determinants, and potential mechanisms of intervention effects to optimize intervention components and implementation strategies for future scale-up, if effective. The specific aims are to:

Specific Aim 1: Test the effectiveness of SPI and TCBT-S for decreasing suicidal behaviors, compared to Enhanced Usual Care (EUC). Using a three-arm parallel cluster RCT the investigators will randomize 7 secondary schools each to EUC, SPI, and TCBT-S (21 schools total) to evaluate effects on suicidal behaviors (primary) and suicidal ideation/depressive symptoms (secondary). EUC will involve screening and active referral to government youth friendly mental health service programs. Exploratory analyses will examine mechanisms of intervention effects.

Specific Aim 2: Assess implementation outcomes and determinants (barriers/facilitators) to EUC, SPI, and TCBT-S implementation using the RE-AIM evaluation framework. RE-AIM domains will be populated separately and compared across arms. The investigators will conduct a sequential quantitative to qualitative explanatory analysis - organized around the Consolidated Framework for Implementation Research - among individuals and clusters with highest/lowest effectiveness/implementation outcomes to explore determinants of implementation.

Specific Aim 3: Estimate the cost and cost-effectiveness of SPI and TCBT-S, compared to EUC. The investigators will conduct micro-costing and time-and-motion observation separately for each study arm to estimate incremental costs of implementing each intervention. The investigators will construct a Markov model parameterized with cost and trial outcomes data to project budget impact and cost-effectiveness for scale-up to provincial and national levels.

This proposal is innovative in being one of the first to rigorously test suicide prevention interventions among African adolescents. In response to the NOSI for Youth Suicide in LMICs (NOT-MH-21-090), this project proposes to test "prevention strategies to reduce suicide risk and promote resilience among young people aged 10-24 years in LMICs". Specifically, this study "integrates suicide prevention strategies within existing community-level platforms such as school/university-based programs" and includes analyses to "determine how to improve fidelity of implementation and economic evaluation of suicide prevention programs for young people". If effective, SPI or TCBT-S have a large potential to be rapidly scaled up to safeguard youth mental health in Mozambique and other similar LMICs.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for suicide risk screening:

1. Youth enrolled in a secondary school in Sofala Province that is located within 30 minutes of a health facility that hosts both an urgent care and mental health department.
2. Youth enrolled in 9th and/or 10th and/or 11th grade.
3. Legal guardian has provided consent to participate if under 18 or if youth is age 18 or older and has provided consent to participate.
4. Youth has assented to participation.

Inclusion criteria for trial participation and allocation to study arm:

1. Youth expresses active suicidal ideation on the Columbia Suicide Severity Rating Scale (C-SSRS).

Exclusion Criteria:

1. Youth and/or guardian has not provided consent to participate, or responsible party is unable to provide informed consent.
2. Youth is not enrolled in a participating secondary school.
3. Youth declines to assent.
4. Youth is a ward of the State or any other agency, institution, or entity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Suicidal Behavior | 6-months post intervention
  As reported on the Columbia Suicide Severity Rating Scale. The responses of the C-SSRS tool are yes or no options that indicate the user's level of risk as low, moderate or high risk of suicide.

SECONDARY OUTCOMES:
Suicidal Behavior - Supplementary analysis of primary outcome | 3-months post intervention
  As reported on the Columbia Suicide Severity Rating Scale. The responses of the C-SSRS tool are yes or no options that indicate the user's level of risk as low, moderate or high risk of suicide.
Suicidal Ideation | 3-, 6-, 12-, and 24-months post intervention
  As reported on the Columbia Suicide Severity Rating Scale. The responses of the C-SSRS tool are yes or no options that indicate the user's level of risk as low, moderate or high risk of suicide.
Depressive Symptoms | 3-, 6-, 12-, and 24-months post intervention
  Depressive symptoms as measured on the Patient Health Questionnaire 9 - MZ, the scoring range is 0-27 with higher scores indicative of more severe symptoms
Suicidal Behavior - Maintenance Indicators | 12-, and 24-months post intervention
  As reported on the Columbia Suicide Severity Rating Scale. The responses of the C-SSRS tool are yes or no options that indicate the user's level of risk as low, moderate or high risk of suicide.

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Wagenaar, PhD, MPH, Principal Investigator — University of Washington
Locations (7):
- Mozambique (7):
  - 9 Secondary Schools, Beira
  - 1 Secondary School, Caia
  - 1 Secondary School, Cheringoma.
  - 1 Secondary School, Chibabava
  - 4 Secondary Schools, Dondo
  - 1 Secondary School, Maringue
  - 4 Secondary Schools, Nhamatanda

REFERENCES:
- [Derived] Wagenaar BH, Muanido A, Turner M, Lovero KL, Darnell D, Sharma M, Comtois KA, Ramiro I, Cumbe VFJ. Safety planning and transdiagnostic cognitive behavioral therapy for adolescent suicide prevention in Mozambique: study protocol for the SPI/TCBT-S hybrid effectiveness/implementation cluster randomized trial. BMC Psychiatry. 2025 Jul 1;25(1):656. doi: 10.1186/s12888-025-07102-w. PMID 40598126